CLINICAL TRIAL: NCT03513549
Title: A Postmarketing Observational Study to Evaluate the Safety of ADASUVE® (STACCATO® Loxapine for Inhalation) in Patients With Agitation Associated With Schizophrenia or Bipolar I Disorder
Brief Title: Observational Study Evaluating the Safety of ADASUVE® in Agitation Associated With Schizophrenia or Bipolar I Disorder
Status: Suspended | Type: Observational
Why Stopped: Suspended due to low patient enrollment resulting from low commercial usage of Adasuve. Study continuation is impractical. Alexza has been in discussions with FDA on this matter.
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Other Study IDs: TV571-CNS-40036
Record Dates: First submitted 2018-04-11; First posted 2018-05-01 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Agitation,Psychomotor
Keywords: Agitation; Schizophrenia; Bipolar I disorder
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia | interventions — Loxapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Loxapine 10 MG: ADASUVE (loxapine) inhalation powder in a 10-milligram (mg) single-use oral inhaler. One dose in a 24-hour period.
  Interventions: Drug: Loxapine 10 MG

INTERVENTIONS:
Drug: Loxapine 10 MG
  Other Names: ADASUVE (loxapine) inhalation powder, NDA 022549

SUMMARY:
This postmarketing observational study will evaluate the safety of ADASUVE® in treating patients with agitation associated with schizophrenia or bipolar I disorder.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study conducted to evaluate the safety of ADASUVE treatment when used in real-world clinical setting in patients with agitation associated with schizophrenia or bipolar I disorder.

The primary objective of the study is to assess the safety of ADASUVE treatment in real-world clinical settings.

The secondary objective of the study is to describe the characteristics of patients, including demographic and baseline characteristics, after administration of ADASUVE treatment in real-world clinical settings.

The study population will consist of a non-randomized cohort of approximately 10000 adult men and women who have agitation associated with schizophrenia or bipolar I disorder (naïve and non-naïve to ADASUVE treatment).

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study if they meet all of the following criteria:

1. The patient is a man or woman who is 18 years of age or older at time of enrollment.
2. The patient is receiving ADASUVE for agitation in a medical or psychiatric emergency setting or in a psychiatric inpatient setting. (Note: Patients with a prior history of treatment with ADASUVE may also be included in the study.)
3. The patient (or caregiver or legally authorized representative) is willing and able to provide written informed consent (and assent, where applicable) after administration of ADASUVE treatment.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a non-randomized cohort of approximately 10000 adult men and women who have agitation associated with schizophrenia or bipolar I disorder (naïve and non-naïve to ADASUVE treatment), as determined by the treating health care provider, and who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-11-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Evaluating frequency and nature of adverse events, serious adverse events and respiratory adverse events of special interest (AESIs) after administration of ADASUVE treatment in real-world clinical settings | 24 hours
  Safety will be assessed by evaluating adverse events, serious adverse events, and respiratory AESIs within the study follow-up period after administration of ADASUVE treatment in real-world clinical settings.

SECONDARY OUTCOMES:
Patient demographics | 24 hours
  The secondary measure of this study is patient characteristics, including demographic characteristics, after administration of ADASUVE treatment in real-world clinical settings.
Patient baseline characteristics - medical history | 24 hours
  The secondary measure of this study is patient characteristics, including baseline characteristic of medical history, after administration of ADASUVE treatment in real-world clinical settings.
Patient baseline characteristics - prior medications | 24 hours
  The secondary measure of this study is patient characteristics, including baseline characteristic of prior medications, after administration of ADASUVE treatment in real-world clinical settings.

OTHER OUTCOMES:
Exploratory objective - patient treatment satisfaction | 24 hours
  The exploratory objective of the study is to assess patient perception of effectiveness (ranging from extremely dissatisfied to extremely satisfied), convenience (ranging from extremely inconvenient to extremely convenient), and overall satisfaction (ranging from extremely dissatisfied to extremely satisfied) using a modified Treatment Satisfaction Questionnaire for Medication (TSQM) after administration of ADASUVE treatment in real-world clinical settings. The TSQM is a modified version of the original TSQM version 1.4, a widely used generic measure to assess treatment satisfaction with medication. Scores range from 0 to 100, with higher scores representing higher satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutical Research Associates, Inc, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No